CLINICAL TRIAL: NCT02551302
Title: "Efficacy of Hybrid Systems ("Topping Off") Versus Rigid Spinal Fusion in Lumbar Fusion Surgery: A Dual-center, Prospective, Randomized Pilot Study ("CD Horizon BalanC")"
Acronym: BalanC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cologne (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. Jan Siewe, Dr.med., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ortho-6-2015
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Spine Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLIF (Other): The control group will receive a monosegmental posterior lumbar spine fusion with an intervertebral cage (PLIF).
  Interventions: Device: Solera™ Medtronic
- Hybrid system (PLIF + flexible pedicle screw system above the (Other): The intervention group will receive a hybrid system with a PLIF and a flexible pedicle screw system above the fusion.
  Interventions: Device: CD HORIZON BalanC™ Medtronic

INTERVENTIONS:
Device: Solera™ Medtronic — The control group will receive a monosegmental posterior lumbar spine fusion with an intervertebral cage (PLIF). Solera™ Medtronic
  Arms: PLIF
Device: CD HORIZON BalanC™ Medtronic — The intervention group will receive a hybrid system with a PLIF and a flexible pedicle screw system above the fusion. Surgery will be performed with the following devices:
  CD HORIZON BalanC™ Medtronic
  Arms: Hybrid system (PLIF + flexible pedicle screw system above the

SUMMARY:
Effectiveness of hybrid systems ("topping off") compared to rigid spondylodesis in fusion surgery of the lumbar spine: A prospective, randomized, bicentric pilot study ("CD HORIZON BalanC™)

DETAILED DESCRIPTION:
Posterior spondylodesis and monosegmental intervertebral cage plus flexible spondylodesis of the superiorly adjacent segment (CD HORIZON BalanC™ Manufacturer: Medtronic)

Control:

Posterior spondylodesis and monosegmental intervertebral cage

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Legal capacity
* Age ≥ 30 years
* Indication for monosegmental lumbar spine fusion (PLIF or "topping-off ") L2-S1 with osteochondrosis Modic grades I-III [20][21][22] or spondylolisthesis Meyerding grades I-III.
* Radiologic signs of degeneration in the adjacent segment of the intended fusion without signs of instability

Exclusion Criteria:

* Motor deficit
* Cauda equina syndrome
* Previous surgical intervention of the lumbar spine
* Relevant peripheral neuropathy
* Acute denervation subsequent to a radiculopathy
* Scoliosis with Cobb angle greater than 25°
* Spondylolisthesis > Meyerding grade III
* Radiologic signs of degeneration in the adjacent segment of the intended fusion with signs of instability (for definition, see inclusion criteria)
* No radiologic signs of degeneration in the adjacent segment of the intended fusion (for definition, see inclusion criteria)
* Radiologic signs of degeneration in the adjacent segment of the intended fusion with >Fujiwara grade II [15] or >Pfirrmann grade IV [14]
* Signs of instability in any lumbar spine segment other than that undergoing fusion
* General contraindication for elective lumbar spine surgery
* Pathologic fracture
* Osteoporosis with pathologic fracture
* Active systemic infection
* Rheumatic disease
* Disease of bone metabolism (e.g. Paget's Disease)
* Bone metastasis
* Local infection focus lumbar spine
* Seizure disorder
* Chronic ischemia Fontaine classification IIb-IV
* Severe heart insufficiency (NYHA III-IV)
* Blood coagulation disorder or blood thinning therapy
* Cortisone intake more than one month in the last 12 months before randomization
* Simultaneous participation in another clinical trial in the 30 days before randomization
* Known allergy or intolerance to the implants
* Dependency on investigator
* Lack of familiarity with the German language
* Placement in an institution by governmental or juridical advice
* Absent legal capacity
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the subscores of physical pain and physical function in the ODI Questionaire | Baseline to 6 month

SECONDARY OUTCOMES:
MCS and individual dimensions and subscales of the SF-36™ | 60 Month

CONTACTS AND LOCATIONS:
Overall Officials: Jan Siewe, Dr.med., Principal Investigator — University Hospital Cologne